CLINICAL TRIAL: NCT05766085
Title: Cortisol Secretion, Sensitivity and Activity and Hypertension
Acronym: PRECOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 05C921
Record Dates: First submitted 2023-02-27; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Hypercortisolism; Arterial Hypertension
Keywords: hypertension; hidden hypercortisolism; hypercortisolism; cortisol sensitivity
MeSH Terms: conditions — Cushing Syndrome; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypertension: Those patients suffering from arterial hypertension
  Interventions: Diagnostic Test: Dexamethasone suppression test
- no hypertension: Those patients without arterial hypertension
  Interventions: Diagnostic Test: Dexamethasone suppression test

INTERVENTIONS:
Diagnostic Test: Dexamethasone suppression test — Determination of cortisol levels at 9.00 am after taking 1 mg of dexamethasone the previous evening at 11.00 pm (1mg DST)

SUMMARY:
The goal of this observational study is to evaluate, between patients with arterial hypertension and non hypertensive control group,

* the prevalence of hidden hypercortisolism
* the relationship between organ damage and oxidative stress level, cortisol secretion degree, sensitivity and peripheral activity

ELIGIBILITY:
Inclusion Criteria:

* Hypertension group: arterial hypertension
* No hypertension group: absence of arterial hypertension

Exclusion Criteria:

* body mass index (BMI) >30 kg/m2
* active smoking (>20 cigarettes/day)
* pregnancy/lactation
* hypertension associated with family history of hypertension and cerebrovascular events before 40 years of age
* sleep apnea
* hypertension appearance in pre-pubertal age
* hypokalemia
* hypertension in the setting of an incidental adrenal mass
* classic signs and symptoms of hypercortisolism (lunar facies, striae, hypertrichosis, skin atrophy, hump)
* proven endocrine hypertension (pheochromocytoma, hyperaldosteronism, hyperparathyroidism, acromegaly, hyperthyroidism)
* renovascular hypertension
* diseases or conditions associated with increased activity of the hypothalamic-pituitary- adrenal axis and/or oxidative stress, such as type 2 diabetes, rheumatoid arthritis, severe rheumatic/autoimmune diseases, severe hematological diseases, alcoholism, depressive syndrome, chronic renal failure (GFR <45 ml/min), severe hypovitaminosis D (25OHvitaminD <10 ng/dL)
* therapies that interfere with the activity of the HPA axis (i.e. glucocorticoids, antidepressants).

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertension group: patients with hypertension referred to the cardiology clinics of Istituto Auxologico Italiano, Milan No hypertension group: patients without hypertension referred to endocrinology clinics of Istituto Auxologico Italiano for other diseases (e.g. euthyroid nodular goiter or chronic lymphocytic euthyroid thyroiditis)
Sampling Method: Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hidden hypercortisolism (HidHyCo) | At baseline
  The presence of HidHyCo will be evaluated through the determination of cortisol levels at 9.00 am after taking 1 mg of dexamethasone the previous evening at 11.00 pm (1mgDST). In case of 1mgDST >1.8 µg/dL the patient will repeat the test and, if the result is confirmed, the patients is considered to have HidHyCo.

SECONDARY OUTCOMES:
Evaluation of organ damage | At baseline
  Organ damage will be assessed by performing echocardiography, carotid echo-doppler (arterial stiffness) and microalbuminuria evaluation, which assess hypertensive heart disease, macro-angiopathy and hypertensive nephropathy, respectively
Evaluation of oxidative stress level | At baseline
  The determination of the degree of oxidative stress will be carried out in all patients by evaluating the enzymatic activity of dipeptidyl peptidase 3 (DPP3) in the serum
Evaluation of cortisol secretion degree | At baseline
  The cortisol secretion will be evaluated by measuring morning plasma ACTH and serum cortisol, 24-hour urinary free cortisol, serum cortisol at 09:00 after the administration of
  1 mg dexamethasone at 11 PM on the previous day
Evaluation of glucocorticoid sensitivity | At baseline
  In all subjects, genotyping of the N363S, BclI, ER22/23EK polymorphisms of the GR gene and of the polymorphisms will be performed
Evaluation of glucocorticoid peripheral activity | At baseline
  Urinary free cortisol and urinary free cortisone will be measured in all subjects; their ratio will be used as measure of glucocorticoid peripheral activity

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Aresta, MD, Principal Investigator — Istituto Auxologico Italiano IRCCS
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, MI, Italy